CLINICAL TRIAL: NCT01087957
Title: Randomized Trial of the Innovative Neurotronics WalkAide Compared to Conventional Ankle-Foot Orthosis (AFO) in Stroke Patients (INSTRIDE)
Brief Title: WalkAide Compared to Ankle-Foot Orthosis (AFO) in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovative Neurotronics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INSTRIDE
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ankle-Foot Orthosis (AFO) (Active Comparator): Comparison of WalkAide device against Ankle-Foot Orthosis (AFO)
  Interventions: Other: Ankle-Foot Orthosis (AFO)
- WalkAide (Active Comparator): Comparison of WalkAide device against Ankle-Foot Orthosis (AFO)
  Interventions: Device: WalkAide

INTERVENTIONS:
Device: WalkAide — Comparison of WalkAide device against Ankle-Foot Orthosis (AFO)
  Arms: WalkAide
Other: Ankle-Foot Orthosis (AFO) — Comparison of WalkAide device against Ankle-Foot Orthosis (AFO)
  Arms: Ankle-Foot Orthosis (AFO)

SUMMARY:
To establish equivalence or incremental benefit to standard of care Ankle-Foot Orthosis (AFO) for patients with foot drop due to stroke, and to assess the functional improvement of ambulation and improved activities of daily living.

DETAILED DESCRIPTION:
This is a pivotal un-blinded, randomized, controlled trial with parallel group therapeutic intervention versus control of standard of care (AFO).

ELIGIBILITY:
Inclusion Criteria:

* Patient history of stroke (ischemic and/or hemorrhagic).
* Patient is at least 6 months post stroke.
* Patient has hemiplegia/hemiparesis.
* Patient has inadequate dorsiflexion during swing phase of gait, resulting in inadequate limb clearance.
* Patient is not currently using Functional Electrical Stimulation for the treatment of footdrop.
* Patient is a minimum of 30 days post inpatient or outpatient stroke, cardiac, pulmonary, or physical rehabilitation on the lower extremity.
* Patient is a minimum of 90 days post major orthopedic surgery (i.e. hip, knee, and/or ankle joint replacement).
* Patient is a minimum of 90 days post myocardial infarction.
* Patient is a minimum of 90 days post stenting procedure (i.e. peripheral, cardiac, carotid, and/or renal).
* Patient is a minimum of 6 months post CABG or cardiac valve procedure.
* Patient is able to walk at least 10 meters with or without an assist device (excluding an AFO or WalkAide device).
* Patient has an initial gait speed > 0.0 m/s and < 0.8 m/s.
* Patient has a positive response to peroneal nerve stimulation testing, resulting adequate dorsiflexion of the ankle.
* Patient has adequate cognitive function to permit reliable completion of evaluation instruments and to correctly use the therapeutic interventions as determined by a Mini-Mental Status test score >17 within 30 days prior to enrollment.
* Patient has completed a full neurological assessment within 30 days prior to enrollment.
* Patient is eligible for Medicare or Medicare Choice/Advantage benefits at the time of enrollment
* Patient is able and willing to comply with study procedures, including follow-up requirements.
* Patient is able and willing to give written informed consent.

Exclusion Criteria

* Patient is less than 6-months post stroke.
* Patient has inadequate cognitive function to permit reliable completion of evaluation instruments and to correctly use the therapeutic interventions as determined by a Mini-Mental Status test score < 17 within 30 days prior to enrollment.
* Patient has ankle joint instability other than foot drop.
* Patient is less than 30 days post inpatient or outpatient: stroke, cardiac, pulmonary, or any type of physical rehabilitation on the lower extremity at time of enrollment.
* Patient has need for an AFO for stance control of the foot, ankle and/or knee.
* Patient has an initial gait speed of 0.8 m/s or greater classified as a full community walker (independent in all home and community activities).
* Patient is not able to safely clear toes in swing phase on the involved lower extremity, defined as >-5° plantar flexion, with the device determined at fitting visit.
* Patient has been diagnosed with peripheral neuropathy and symptoms obstruct or limit ambulation or participation in study procedures.
* Patient has been diagnosed with significant peripheral vascular disease accompanied by lower extremity ulceration and/or disabling claudication.
* Patient has underlying condition(s) that would limit study participation such as severe hypertonicity resulting in the need for more involved orthotic strategies or excessive dysesthetic pain secondary to neurological involvement.
* Patient has moderate to very severe COPD, as defined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD).
* Patient is NYHA Class III or IV.
* Patient has malignant skin lesion below the knee on the affected lower extremity.
* Patient has history of seizure disorder and on seizure medications.
* Patient has aphasia, defined as incapacity to verbalize commands.
* Patient has Beck Depression Index score of > 29 indicating severe depression.
* Patient has a life expectancy less than 12 months.
* Patient has existing electrical stimulation devices (ICD, Pacemaker, Spinal Stimulation, TENS).
* Patient is less than 6 months free from Botulinum Toxin (Botox) injection in the lower extremity.
* Patient has baclofen pump with unstable dosing in the last 3 months.
* Patient is unable or unwilling to comply with study procedures, including follow-up requirements.
* Patient is participating in another clinical trial that, according to the Principal Investigator, is likely to affect study outcome or confound results.
* Patient is unable or unwilling to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Bethoux, M.D., Principal Investigator — The Cleveland Clinic
Locations (29):
- United States (29):
  - The Loma Linda University Medical Center, Loma Linda, California
  - The Los Angeles VA, Los Angeles, California
  - Casa Colina Centers for Rehabilitation, Pomona, California
  - The San Francisco VA Medical Center, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - Halifax Hospital, Daytona Beach, Florida
  - Florida Hospital NORI, Orlando, Florida
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Marianjoy Rehabilitation, Wheaton, Illinois
  - Cardinal Hill Rehabilitation, Lexington, Kentucky
  - St. Mary's of Michigan, Saginaw, Michigan
  - University of Minnesota Twin-Cities, Minneapolis, Minnesota
  - Madonna Rehabilitation Hospital, Lincoln, Nebraska
  - Kessler Foundation Research Center, West Orange, New Jersey
  - United Healthcare, Johnson City, New York
  - South Shore Neurologic Associates, Patchogue, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Health Research Inc./Helen Hayes Hospital, West Haverstraw, New York
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - FirstHealth of the Carolinas, Pinehurst, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Magee Rehabilitation Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. David's Rehabilitation Hospital, Austin, Texas
  - The Dallas VA, Dallas, Texas
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Result] Bethoux F, Rogers HL, Nolan KJ, Abrams GM, Annaswamy TM, Brandstater M, Browne B, Burnfield JM, Feng W, Freed MJ, Geis C, Greenberg J, Gudesblatt M, Ikramuddin F, Jayaraman A, Kautz SA, Lutsep HL, Madhavan S, Meilahn J, Pease WS, Rao N, Seetharama S, Sethi P, Turk MA, Wallis RA, Kufta C. The effects of peroneal nerve functional electrical stimulation versus ankle-foot orthosis in patients with chronic stroke: a randomized controlled trial. Neurorehabil Neural Repair. 2014 Sep;28(7):688-97. doi: 10.1177/1545968314521007. Epub 2014 Feb 13. PMID 24526708
- [Derived] Bethoux F, Rogers HL, Nolan KJ, Abrams GM, Annaswamy T, Brandstater M, Browne B, Burnfield JM, Feng W, Freed MJ, Geis C, Greenberg J, Gudesblatt M, Ikramuddin F, Jayaraman A, Kautz SA, Lutsep HL, Madhavan S, Meilahn J, Pease WS, Rao N, Seetharama S, Sethi P, Turk MA, Wallis RA, Kufta C. Long-Term Follow-up to a Randomized Controlled Trial Comparing Peroneal Nerve Functional Electrical Stimulation to an Ankle Foot Orthosis for Patients With Chronic Stroke. Neurorehabil Neural Repair. 2015 Nov-Dec;29(10):911-22. doi: 10.1177/1545968315570325. Epub 2015 Feb 4. PMID 25653225

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Started | 253 | 242
Completed | 212 | 187
Not Completed | 41 | 55
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 3 | 4
Not completed — Protocol Violation | 13 | 25
Not completed — Withdrawal by Subject | 18 | 15
Not completed — Physician Decision | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide | Total
Number analyzed (Participants) | 253 | 242 | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.30 (12.01) | 63.87 (11.33) | 64.09 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 95 | 191
  Male | 157 | 147 | 304
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 55 | 55 | 110
  White | 187 | 177 | 364
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 8 | 13
Time Post Onset of Stroke [Mean (Standard Deviation); unit: years] | 6.86 (6.64) | 6.90 (6.43) | 6.88 (6.53)
Initial Gait Speed [Mean (Standard Deviation); unit: meters/second] | .487 (.21) | .449 (.22) | .47 (.21)
Mini Mental Status Exam [Mean (Standard Deviation); unit: units on a scale] — The Mini Mental Status is a measure of cognitive function with a total possible score of 30 points. Any score greater than or equal to 27 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-24 points) cognitive impairment
  units on a scale | 27.49 (2.83) | 27.62 (2.44) | 27.54 (2.65)
Beck Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression inventory is a 21-question multiple-choice self-report inventory used for measuring the severity of depression. Each of the 21 questions is scored on a scale value of 0 to 3. Total score thresholds recommendations are as follows: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; and 29-63: severe depression. Higher total scores indicate more severe depressive symptoms.
  units on a scale | 8.08 (6.58) | 7.98 (6.32) | 8.05 (6.45)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meters squared] | 29.21 (5.08) | 27.98 (4.93) | 28.61 (5.04)

OUTCOME MEASURES:

1. Primary Outcome: Gait Velocity
Description: Improved ambulation status, specific to increase in gait velocity (m/s)
Time Frame: 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: m/sec
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
m/sec | .682 (.020) | .635 (.022)

2. Primary Outcome: Stroke Impact Scale (SIS) Composite Score
Description: The SIS Composite score is equal to sum of scores for Mobility, ADL/IADL, and Social Participation domains. The questions for each domain are scored on a scale of 1-5, the higher the score the less the impact of Stroke on that domain question. The Mobility domain has 9 questions with scores ranging from 9 to 45. The ADL/IADL domain has 10 questions with scores ranging from 10-150- and the Social Participation domain has 8 question with a score of 8-40.
Time Frame: 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
points | 172.7 (2.8) | 175.0 (2.7)

3. Primary Outcome: Device Related Serious Adverse Events
Description: The device related serious adverse event (SAE) measure is a count of the incidences of adverse events defined as serious (Incapacitating with inability to do work or usual activities; signs and symptoms may be systemic in nature or require medical evaluation and/or treatment; requiring additional hospitalization or intensive care (prolonged hospitalization) and device related (any AE for which a causal relationship between the event and the presence of the device, or the performance of the device system, is at least a reasonable possibility (i.e., the relationship cannot be excluded).
Time Frame: 6 months
Population: Intention to treat
Measure: Number; unit: number of device related SAEs
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
number of device related SAEs | 2 | 0

4. Secondary Outcome: Six Minute Walk Test
Time Frame: 6 months
Measure: Mean (Standard Error); unit: meters
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
meters | 218.6 (7.6) | 209.2 (8.5)

5. Secondary Outcome: Modified Emory Functional Ambulation Profile Total Score
Description: The Modified Emory Functional Ambulation Profile (mEFAP) is composed of 5 subtasks: (1) 5 meter walk on a hard Floor, (2) 5 meter walk on a carpeted surface, (3) Timed Up & Go (rising from a chair, a 3-meter walk, and return to a seated position), (4) Navigating a Standardized Obstacle Course, and (5) ascending and descending 4 Stairs. Each is a timed task with the score consisting of the number of seconds required to complete the task. Upon completion of the entire data collection session, a total mEFAP score is calculated by adding the score on each subtask.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
seconds | 479.4 (38.3) | 498.0 (32.0)

6. Secondary Outcome: Modified Emory Functional Ambulation Profile Floor Time
Description: The Modified Emory Functional Ambulation Profile (mEFAP) Floor time sub-task is composed a timed 5 meter walk on a hard Floor. The score consists of the number of seconds required to complete the task. The Floor Time sub-task is added to the other 4 sub-tasks to make up the total mEFAP score.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
seconds | 56.0 (8.0) | 52.5 (3.9)

7. Secondary Outcome: Modified Emory Functional Ambulation Profile Carpet Time
Description: The Modified Emory Functional Ambulation Profile (mEFAP) Carpet time sub-task is composed of a 5 meter walk on a carpeted surface with the score consisting of the number of seconds required to complete the task. The score on the Carpet time sub-task is added to the other 4 sub-tasks to calculate the total mEFAP score .
Time Frame: 6 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
seconds | 56.1 (6.6) | 57.1 (4.4)

8. Secondary Outcome: Modified Emory Functional Ambulation Profile Timed up and Go
Description: The Modified Emory Functional Ambulation Profile (mEFAP) Timed up and Go subtask is composed of rising from a chair, walking 3-meters, and returning to a seated position with the score consisting of the number of seconds required to complete the task. The Timed up and Go subtask is added to the other 4 sub-task scores to calculate the total mEFAP score.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
seconds | 131.0 (14.7) | 126.9 (9.4)

9. Secondary Outcome: Modified Emory Functional Ambulation Profile Obstacle Course
Description: The Modified Emory Functional Ambulation Profile (mEFAP) Obstacle course sub-task is composed navigating a Standardized Obstacle Course with the score consisting of the number of seconds required to complete the task. The obstacle course sub-task is added to the other 4 sub-tasks to calculate the total mEFAP score.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
seconds | 169.8 (11.8) | 182.2 (14.8)

10. Secondary Outcome: Modified Emory Functional Ambulation Profile Stair Time
Description: The Modified Emory Functional Ambulation Profile (mEFAP) Stair time sub-task is composed of ascending and descending 4 Stairs with the score consisting of the number of seconds required to complete the task. The Stair time sub-task score is added to the other 4 subtask scores to calculate the total mEFAP score .
Time Frame: 6 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
seconds | 66.4 (5.3) | 79.3 (5.9)

11. Secondary Outcome: Berg Balance Scale
Description: The Berg Balance Assessment is a 14 item scale designed to measure balance in adults in a clinical setting. Each item is scored on a scale of 0-4 with a score of 0 indicating the most difficulty with the balance task. A score from 0 to 20 represents balance impairment, 21 to 40 represents acceptable balance, and 41-56 represents good balance.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Number analyzed (Participants) | 253 | 242
units on a scale | 44.7 (0.8) | 44.9 (0.6)

ADVERSE EVENTS:
Arm/Group | Ankle-Foot Orthosis (AFO) | WalkAide
Serious Adverse Events (participants affected / at risk) | 17/253 | 18/242
Other Adverse Events (participants affected / at risk) | 146/253 | 162/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ankle-Foot Orthosis (AFO) (N=253) | WalkAide (N=242)
Fall (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Death (Nervous system disorders) | 2 (2) | 1 (1)
Death (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 3 (5) | 5 (9)
Back surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
TIA or CVA (Nervous system disorders) | 3 (4) | 5 (6)
Renal failure/infection (Renal and urinary disorders) | 1 (2) | 3 (5)
Hospitilization GI disorder (Gastrointestinal disorders) | 4 (4) | 0 (0)
Hospitilized for abnormal Blood Sugar level (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ankle-Foot Orthosis (AFO) (N=253) | WalkAide (N=242)
Falls (Musculoskeletal and connective tissue disorders) | 89 (173) | 99 (173)
Pain in back or Lower Extremity (Musculoskeletal and connective tissue disorders) | 30 (55) | 26 (36)
Fatigue/Muscle weakness (Pregnancy, puerperium and perinatal conditions) | 9 (18) | 3 (4)
Other medical conditions (Surgical and medical procedures) | 65 (166) | 70 (149) — Various events involving multiple systems
Skin Irritation (Skin and subcutaneous tissue disorders) | 10 (10) | 29 (34)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 11 (15) | 12 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
(b) Publication- Investigator and Institution agree not to publish the results of the Trial until after the conclusion of the Trial. Investigator agrees to submit to Sponsor copies of any proposed publication at least sixty (60) calendar days in advance of dissemination. Sponsor agrees to review and comment in a timely manner after receipt . All proprietary and/or confidential information of Sponsor must be removed from the Proposed Publication.